CLINICAL TRIAL: NCT07073443
Title: Evaluation of the Effect of Memory-based Reminiscence Therapy on Cognitive Status, Psychological Flexibility and Cognitive Flexibility in Older People With Dementia
Brief Title: Evaluation of the Effect of Memory-based Reminiscence Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaraş İstiklal University (Other)
Responsible Party: Principal Investigator, Pinar Harmanci, Associate Professor, Kahramanmaraş İstiklal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstiklalU-Harmanci-002
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Memory, Short-Term
Keywords: Memory therapy; memory; cognitive state; psychological flexibility; cognitive flexibility
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memory Therapy Group (Experimental): The intervention group of elderly individuals underwent 10 sessions of Memory Therapy, with two sessions per week over a period of five weeks. The sessions were planned to last an average of 45 minutes. During the 10 sessions, Memory-Based Reminiscence Therapy was applied to the intervention group using reminiscence phenomena and verbal reminders were provided in repetitive narratives.
  Interventions: Behavioral: Experimental: Memory Therapy Group
- Control group (No Intervention): No intervention was made for individuals in this group.

INTERVENTIONS:
Behavioral: Experimental: Memory Therapy Group — Evaluation of the Effect of Memory-Based Recall Therapy on the Cognitive Status, Psychological Flexibility, and Cognitive Flexibility of Elderly Individuals Diagnosed with Dementia
  Arms: Memory Therapy Group

SUMMARY:
The main objective of this study is to examine the effects of memory-based recall therapy applied to elderly adults diagnosed with Stage 0, 1, and 2 dementia on their mental state, psychological flexibility, and cognitive flexibility.

The original flow plan created in the study is not found in the literature. Therefore, presenting the effects of memory-based recall on cognition in the literature may demonstrate that the contents of classical recall therapy can also be effectively restructured with cognitive effects. From this perspective, the aim is to make recommendations for "advanced psychiatric nursing practices."

Research Hypotheses:

H0: Memory-based recall therapy has no effect on mental state, psychological flexibility, and cognitive flexibility in individuals with early-stage dementia.

H1: Memory-based Recall Therapy has an effect on mental state, psychological flexibility, and cognitive flexibility in individuals with early-stage dementia.

DETAILED DESCRIPTION:
Memory therapy is very important for elderly people with declining cognitive functions, as it can stimulate various senses such as touch, taste, and smell. Materials that facilitate recall can be used in therapy. Physical objects that the elderly can look at and touch provide the patient with additional sources of information, draw their attention to the topics being discussed, and refocus them. In addition, Memory Therapy is a good method for recalling memories and movements that are not readily available or otherwise inaccessible.

The study will be conducted with elderly individuals who have applied to community health centers based in Kahramanmaraş or to the neurology and psychiatry departments of tertiary hospitals. The sample size of 573 was determined based on data obtained from outpatient clinics and community health units (diagnosis sites). At least 114 participants must be reached. Data collection will utilize the Demographic Information Form, Standardized Mini Mental Test (SMMT), Psychological Flexibility Scale, and Cognitive Flexibility Scale. The data will be collected by the researcher in two stages, pre-test and post-test, from all elderly individuals through face-to-face interviews. The elderly in the intervention group will undergo 10 sessions of Memory Therapy, twice a week for five weeks. The sessions will be planned to last an average of 45 minutes. During the 10 sessions of Memory-Based Recall Therapy applied to the intervention group, memory-enhancing phenomena will be used, and verbal reminders will be provided during repeated narratives.

ELIGIBILITY:
Inclusion Criteria:

* Receiving outpatient treatment for dementia from the relevant departments of hospitals
* At the time of the interviews, the doctor must have diagnosed mild dementia. (Stages 0, 1, and 2)
* No problems with understanding or speaking Turkish
* Being literate
* Being in the 65 and older age group
* No other psychiatric or neurological disorders

Exclusion Criteria:

* Not having been diagnosed with dementia during the study
* Having other chronic cognitive and psychiatric illnesses
* Being in an advanced stage of dementia
* Those who withdrew from the study during the interview or refused to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Standardized Mini Mental Test | 0 weeks
  The original Mini Mental Test developed by Folstein et al. (1975) and the standardized version created by Molloy and Standish (1997) are easy to administer and provide information about the degree of cognitive impairment. The lowest possible score on the scale is "0," and the highest possible score is "30." Based on the scores obtained, 0-12 points indicate "severe" cognitive impairment, 13-22 points indicate "moderate" cognitive impairment, 23-24 points indicate 'mild' cognitive impairment, and 25-30 points indicate "no cognitive impairment."
Standardized Mini Mental Test | 5 weeks
  The original Mini Mental Test developed by Folstein et al. (1975) and the standardized version created by Molloy and Standish (1997) are easy to administer and provide information about the degree of cognitive impairment. The lowest possible score on the scale is "0," and the highest possible score is "30." Based on the scores obtained, 0-12 points indicate "severe" cognitive impairment, 13-22 points indicate "moderate" cognitive impairment, 23-24 points indicate 'mild' cognitive impairment, and 25-30 points indicate "no cognitive impairment."
Psychological Flexibility Scale | 0 weeks
  The scale developed by Francis et al. in 2016 was translated into Turkish by Karakuş and Akbay (2020) and underwent validity and reliability testing. The scale consists of 28 items and is a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). The Cronbach's alpha value for the total scale in the Turkish validity and reliability study was 0.79, 0.84 for the values and values-based behavior subscale, 0.60 for the "being in the moment" subscale, 0.72 for the 'acceptance' subscale, 0.73 for the "contextual self" subscale, and 0.59 for the "separation" subscale.
Psychological Flexibility Scale | 5 weeks
  The scale developed by Francis et al. in 2016 was translated into Turkish by Karakuş and Akbay (2020) and underwent validity and reliability testing. The scale consists of 28 items and is a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). The Cronbach's alpha value for the total scale in the Turkish validity and reliability study was 0.79, 0.84 for the values and values-based behavior subscale, 0.60 for the "being in the moment" subscale, 0.72 for the 'acceptance' subscale, 0.73 for the "contextual self" subscale, and 0.59 for the "separation" subscale.
Cognitive Flexibility Inventory | 0 weeks
  Cognitive Flexibility Inventory (CFI) The Cognitive Flexibility Inventory (CFI) is a short self-report scale developed to measure cognitive flexibility, which is necessary for individuals to adapt to changing environmental stimuli and replace maladaptive thoughts with more balanced and adaptive ones. The scale yields three distinct types of scores: a total cognitive flexibility score, an "alternatives" subscale score, and a "control" subscale score. Higher scores indicate greater cognitive flexibility. The Cronbach's alpha coefficient for the entire scale was found to be .90.
Cognitive Flexibility Inventory | 5 weeks
  Cognitive Flexibility Inventory (CFI) The Cognitive Flexibility Inventory (CFI) is a short self-report scale developed to measure cognitive flexibility, which is necessary for individuals to adapt to changing environmental stimuli and replace maladaptive thoughts with more balanced and adaptive ones. The scale yields three distinct types of scores: a total cognitive flexibility score, an "alternatives" subscale score, and a "control" subscale score. Higher scores indicate greater cognitive flexibility. The Cronbach's alpha coefficient for the entire scale was found to be .90.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Istiklal Universty, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No